CLINICAL TRIAL: NCT04797598
Title: Effects of Virtual Reality and Cyclic Training on Balance in Sub-acute Stroke
Brief Title: Effects of Virtual Reality and Cyclic Training on Balance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/LHR/20/2054 Qandil Akram
Record Dates: First submitted 2021-03-10; First posted 2021-03-15 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Stroke, Acute
Keywords: Stroke; Virtual Reality; Cyclic Training; Active Video gaming
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Its a randomized control trial, used to compare the effects of virtual reality and cyclic training on balance in sub-acute stroke patients. Subjects with sub-acute stroke meeting the predetermined inclusion and exclusion criteria will be divided into two groups using simple random sampling technique
Who Masked: Participant
Masking Description: Participants will get separate treatment protocols and possible efforts will be put to m ask the both groups about their treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality group (Active Comparator): In this group patients will be treated with virtual reality . This group will receive therapy session for 1 hour, two times in a week and for 12 weeks, total session will be 24. The virtual reality group will receive 30 minutes virtual reality training and 30 minutes conventional treatment.
  Interventions: Other: Virtual reality group
- Cyclic training group (Active Comparator): In this group patients will be treated with cyclic training . This group will receive therapy session for 1 hour, two times in a week and for 12 weeks, total session will be 24. The cyclic training group will receive 30 minutes cyclic training and 30 minutes conventional treatment
  Interventions: Other: Cyclic training group

INTERVENTIONS:
Other: Virtual reality group — This will receive Virtual reality sessions and both group will receive conventional physical therapy as base line treatment
  Arms: Virtual Reality group
Other: Cyclic training group — This will receive cyclic training session. both group will receive conventional physical therapy as base line treatment
  Arms: Cyclic training group

SUMMARY:
Stroke is the third leading cause of functional disability and death in the world. It leads to many problems that affect gait, upper extremity function and balance. In stroke patients balance dysfunction leads to impaired postural control and walking. Because of poor balance fall rate increases in stroke patients. Balance is an important predictor of outcome in stroke rehabilitation. After stroke difficulties in balance control may be caused by multiple factors such as muscle weakness, impaired proprioception, and asymmetry in weight wearing, spasticity and impaired motor control. Different means are used to treat stroke, some conventional treatments along with new adjunct therapies are usual practice for the rehabilitation of the stroke.

Virtual Reality is choice of adjunct therapy now a days and can be used in different ways for the rehabilitation. Virtual Reality or active video gaming proved their role as vital part of the treatment program in pediatric rehabilitation as well as adult rehabilitation program. These programs help the patient to achieve goals for functional and activities of daily living skills.

DETAILED DESCRIPTION:
This study will be a randomized control trial, used to compare the effectiveness of virtual reality and cyclic training on balance in sub-acute stroke patients. Subjects with sub-acute stroke meeting the predetermined inclusion and exclusion criteria will be divided into two groups using simple random sampling technique. Assessment will be done by using berg balance scale (BBS) and time up and go test. Subjects in one group will be treated with Virtual reality and Conventional therapy and in other group Cyclic training and Conventional therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Sub-acute stroke
2. Able to stand for 5 minutes
3. The score of mini mental state examination (MMSE) > 19
4. Male and Females (both genders)
5. Verbal instructions can follow

Exclusion Criteria:

1. Visual and auditory problem unable to hear and see feedback from the video game and problem of vestibular system
2. Spasticity of lower limb
3. Any other medical condition that could affect movement and balance
4. Use of pacemaker, apraxia, epilepsy
5. Psychiatric disorders

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Berg Balance scale | 12 weeks
  this tool is used for assessing change from baseline .14 item scale designed to measure balance among older people with impairment in balance function by assessing the performance of functional tasks.it is a 14 item scale list with each item consisting of a five point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 indicating the highest level of function. BBS have high validity and reliability of 0.98 41 -56= low fall risk 21-40 = medium fall risk 0-20 = high risk
Time up and Go | 12 weeks
  The Timed Up and Go test (TUG) is a simple test used to assess a person's mobility and requires both static and dynamic balance.
  It uses the time that a person takes to rise from a chair, walk three meters, turn around 180 degrees, walk back to the chair, and sit down while turning 180 degrees.
  Interpretation: ≤ 10 seconds = normal. ≤ 20 seconds = good mobility, can go out alone, mobile without gait aid. ≤ 30 seconds = problems, cannot go outside alone, requires gait aid. * A score of ≥ 14 seconds has been shown to indicate high risk of falls.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Asif A Javed, MS, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yang S, Hwang WH, Tsai YC, Liu FK, Hsieh LF, Chern JS. Improving balance skills in patients who had stroke through virtual reality treadmill training. Am J Phys Med Rehabil. 2011 Dec;90(12):969-78. doi: 10.1097/PHM.0b013e3182389fae. PMID 22019971